CLINICAL TRIAL: NCT02500316
Title: Safety and Dose Finding Study of Different MOD-4023 Dose Levels Compared to Daily R-human Growth Hormone (hGH) Therapy in Pre-pubertal Growth Hormone Deficient Children
Brief Title: Long Term Follow up Study of Long-acting hGH (MOD-4023) in Growth Hormone Deficient Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-4-004-OLE; 2011-004553-60 (EudraCT Number)
Record Dates: First submitted 2015-07-12; First posted 2015-07-16 (Estimated); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Growth Hormone Deficiency (GHD)
Keywords: Growth hormone deficiency (GHD); r-hGH; Long-acting
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — MOD-4023

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MOD-4023 (Experimental): Once weekly injection of long acting r-hGH (MOD-4023) provided as a solution for injection containing 20 or 50 mg/mL MOD-4023 in a single patient use, multi-dose, disposable pre-filled pen (PEN).
  Interventions: Drug: MOD-4023

INTERVENTIONS:
Drug: MOD-4023 — Once weekly injection of long acting r-hGH (MOD-4023) provided as a solution for injection containing 20 or 50 mg/mL MOD-4023 in a single patient use, multi-dose, disposable pre-filled pen (PEN).

SUMMARY:
Protocol CP-4-004-OLE (Open Label Extension) is designed as a long-term, open-label extension using single patient use, multi-dose, disposable pre-filled pen.

ELIGIBILITY:
Inclusion Criteria:

Patients who completed the first year of treatment in the main study are allowed to enter the (Long Term) Open Label Extension (OLE) study.

Exclusion Criteria:

1. Children with past or present intracranial tumor growth as confirmed by an MRI scan (with contrast).
2. History of radiation therapy or chemotherapy.
3. Malnourished children defined as:

   1. Serum albumin below the lower limit of normal (LLN) according to the reference ranges of central laboratory;
   2. Serum iron below the lower limit of normal (LLN) according to the reference ranges of central laboratory;
   3. BMI < -2 Standard Deviation for age and sex;
4. Children with psychosocial dwarfism.
5. Children born small for gestational age (SGA - birth weight and/or birth length < -2 SD for gestational age).
6. Presence of anti-hGH antibodies at screening.
7. Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to, chronic diseases like renal insufficiency, spinal cord irradiation, etc.
8. Patients with diabetes mellitus.
9. Patients with impaired fasting sugar (based on WHO; fasting blood sugar >110 mg/dl or 6.1 mmol/l) after repeated blood analysis.
10. Chromosomal abnormalities and medical "syndromes" (Turner's syndrome, Laron syndrome, Noonan syndrome, Prader-Willi Syndrome, Russell-Silver Syndrome, short stature homeobox-containing gene (SHOX) mutations/deletions and skeletal dysplasias), with the exception of septo-optic dysplasia.
11. Closed epiphyses.
12. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids and methylphenidate for attention deficit hyperactivity disorder (ADHD), with the exception of hormone replacement therapies (thyroxine, hydrocortisone, desmopressin (DDAVP))
13. Children requiring glucocorticoid therapy (e.g. asthma) who are taking a dose of greater than 400 µg/d of inhaled budesonide or equivalents for longer than 1 month during a calendar year.
14. Major medical conditions and/or presence of contraindication to r-hGH treatment.
15. Known or suspected HIV-positive patient, or patient with advanced diseases such as AIDS or tuberculosis.
16. Drug, substance, or alcohol abuse.
17. Known hypersensitivity to the components of study medication.
18. Other causes of short stature such as coeliac disease, hypothyroidism and rickets.
19. The patient and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct.
20. Participation in any other trial of an investigational agent within 30 days prior to Screening.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2023-11 (Actual); Study Completion 2023-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Zadik, MD, Principal Investigator — Kaplan Medical Center, Israel
Locations (13):
- Nemours Children's Clinic, Jacksonville, Florida, United States
- 2DKB, Minsk, Belarus
- Children's Hospital "P. A. Kyriakou", Athens, Greece
- Buda Children's Hospital, Budapest, Hungary
- Russia (5):
  - Endocrinology Scientific Centre, Institute of Child Endocrinology, Moscow
  - Russian Medical Academy of Postgraduate Education, Moscow
  - SPGPMA, Saint Petersburg
  - SamGMU, Samara
  - SBEIHPE, Ufa
- Ukraine (4):
  - Donetsk Regional Children Clinical Hospital, Donetsk
  - Institute of Endocrinology, Kiev
  - Ukrainian Scientific Center of Endocrine Surgery Moh of Ukraine, Kiev
  - Odessa Regional Children'S Clinical Hospital, Odesa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MOD-4023
Started | 48
Completed | 21
Not Completed | 27
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 15
Not completed — Final height achieved | 5
Not completed — Due to war activity | 1

BASELINE CHARACTERISTICS:
Population: Full analysis population
Arm/Group | MOD-4023
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.67 (2.122)
Age, Customized [Count of Participants; unit: Participants]
  < 7 years | 25
  ≥ 7 and < 10 years | 13
  ≥ 10 and ≤ 14 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 45
  More than one race | 0
  Unknown or Not Reported | 2
Pubertal Status [Count of Participants; unit: Participants]
  Tanner I (Prepubertal) | 47
  Tanner II (Early puberty) | 1
  Tanner III (Mid puberty) | 0
  Tanner IV (Late puberty) | 0
  Tanner V (Post pubertal) | 0

OUTCOME MEASURES:

1. Primary Outcome: Annualized Height Velocity
Description: A summary of the annualized HV at the end of each year for Periods III/IV (OLE Years 1 - 4) and V (PEN Years 1 - 5).
Time Frame: 8 years
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | MOD-4023
Number analyzed (Participants) | 48
cm/year
  OLE Year 1: number analyzed (Participants) | 46
  OLE Year 1 | 7.99 (1.54)
  OLE Year 2: number analyzed (Participants) | 43
  OLE Year 2 | 7.46 (1.35)
  OLE Year 3: number analyzed (Participants) | 38
  OLE Year 3 | 7.12 (1.66)
  OLE Year 4: number analyzed (Participants) | 1
  OLE Year 4 | 4.63 (NA) — Standard deviation is not applicable for 1 subject
  PEN Year 1: number analyzed (Participants) | 35
  PEN Year 1 | 6.98 (1.89)
  PEN Year 2: number analyzed (Participants) | 31
  PEN Year 2 | 6.37 (2.12)
  PEN Year 3: number analyzed (Participants) | 26
  PEN Year 3 | 5.31 (1.68)
  PEN Year 4: number analyzed (Participants) | 19
  PEN Year 4 | 6.05 (1.74)
  PEN Year 5: number analyzed (Participants) | 2
  PEN Year 5 | 6.31 (0.41)

2. Primary Outcome: Delta Height SDS Every 12 Months
Description: A summary of annual change in height SDS at the end of each year for Periods III/IV (OLE Years 1 - 4) and V (PEN Years 1 - 5). Height SDS (Standard Deviation Score) reflects how an individual's height compares to the average for their age and sex, calculated using Growth Analyzer and based on Switzerland 1989 (Prader) reference. A z-score of 0 indicates a height equal to the population mean, while positive scores indicate above-average heights and negative scores reflect below-average heights.
Time Frame: 8 years
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | MOD-4023
Number analyzed (Participants) | 48
Z-score
  OLE Year 1: number analyzed (Participants) | 46
  OLE Year 1 | 0.57 (0.34)
  OLE Year 2: number analyzed (Participants) | 43
  OLE Year 2 | 0.40 (0.28)
  OLE Year 3: number analyzed (Participants) | 38
  OLE Year 3 | 0.34 (0.28)
  OLE Year 4: number analyzed (Participants) | 1
  OLE Year 4 | 0.09 (NA) — Standard deviation is not applicable for 1 subject
  PEN Year 1: number analyzed (Participants) | 35
  PEN Year 1 | 0.27 (0.25)
  PEN Year 2: number analyzed (Participants) | 31
  PEN Year 2 | 0.21 (0.29)
  PEN Year 3: number analyzed (Participants) | 26
  PEN Year 3 | 0.10 (0.21)
  PEN Year 4: number analyzed (Participants) | 19
  PEN Year 4 | 0.18 (0.34)
  PEN Year 5: number analyzed (Participants) | 2
  PEN Year 5 | 0.07 (0.13)

3. Secondary Outcome: Summary of IGF-1 SDS
Description: A summary of IGF-I SDS at the end of each year for Periods III/IV (OLE Years 1 - 4) and V (PEN Years 1 - 5). IGF-1 SDS (Standard Deviation Score) reflects how an individual's IGF-1 level compares to the average for their age and sex, based on reference values from Bidlingmaier et al. (2014, The Journal of Clinical Endocrinology & Metabolism, 99(5):1712-1721). A z-score of 0 indicates a level equal to the population mean, while positive scores indicate above-average levels and negative scores reflect below-average levels. An IGF-1 SDS below -2 suggests deficiency, whereas a score above +2 is considered elevated. In the study, when IGF-1 SDS exceeded +2, a confirmatory test was performed, and if elevation was confirmed, the dose was reduced by 15%.
Time Frame: 8 years
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | MOD-4023
Number analyzed (Participants) | 48
Z-score
  OLE Year 1: number analyzed (Participants) | 43
  OLE Year 1 | 0.64 (0.96)
  OLE Year 2: number analyzed (Participants) | 41
  OLE Year 2 | 0.65 (1.08)
  OLE Year 3: number analyzed (Participants) | 38
  OLE Year 3 | 1.05 (0.82)
  OLE Year 4: number analyzed (Participants) | 1
  OLE Year 4 | 0.29 (NA) — Standard deviation is not applicable for 1 subject
  PEN Year 1: number analyzed (Participants) | 35
  PEN Year 1 | 1.29 (0.81)
  PEN Year 2: number analyzed (Participants) | 31
  PEN Year 2 | 0.96 (1.15)
  PEN Year 3: number analyzed (Participants) | 26
  PEN Year 3 | 0.86 (0.89)
  PEN Year 4: number analyzed (Participants) | 18
  PEN Year 4 | 1.00 (0.68)
  PEN Year 5: number analyzed (Participants) | 2
  PEN Year 5 | 1.45 (0.33)

ADVERSE EVENTS:
Time Frame: 8 years
Arm/Group | MOD-4023
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 4/48
Other Adverse Events (participants affected / at risk) | 42/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 (N=48)
Gastric disorder (Gastrointestinal disorders) | 1
Thyroid gland abscess (Infections and infestations) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 (N=48)
Upper respiratory tract infection (Infections and infestations) | 13
Bronchitis (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 7
Rhinitis (Infections and infestations) | 7
Tonsillitis (Infections and infestations) | 5
Varicella (Infections and infestations) | 5
Viral upper respiratory tract infection (Infections and infestations) | 5
Ear infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Conjunctivitis (Infections and infestations) | 2
Corona virus infection (Infections and infestations) | 2
Hand-foot-and-mouth disease (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Lower respiratory tract infection viral (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 2
Rotavirus infection (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Scoliosis (Musculoskeletal and connective tissue disorders) | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Delayed puberty (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Secondary hypogonadism (Endocrine disorders) | 2
Pyrexia (General disorders) | 4
Injection site bruising (General disorders) | 2
Injection site erythema (General disorders) | 2
Headache (Nervous system disorders) | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Obesity (Metabolism and nutrition disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Myopia (Eye disorders) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02500316/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT02500316/SAP_001.pdf